CLINICAL TRIAL: NCT02840162
Title: Randomized Study of Pre-Prostatectomy Celecoxib or Placebo
Brief Title: Pre-Prostatectomy Celecoxib or Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug safety concerns
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00001004; HOR-01019-L (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Prostate; Prostate Cancer
Keywords: prostate cancer; NSAIDs; chemoprevention; celecoxib; COX-2 inhibitors
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Celecoxib; Benzenesulfonamides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Active Comparator): Treated patients will receive 4 weeks of celecoxib at 400 mg twice daily by mouth
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Control patients will receive a suitable placebo for 4 weeks, twice daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Selective inhibition of COX-2 without significant cyclooxygenase-1 (COX-1) inhibition
  Other Names: Celebrex; 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]; Benzenesulfonamide
  Arms: Celecoxib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will seek to determine if the downstream effects of cyclooxygenase-2 (COX-2) inhibition suggested by preclinical systems occur in human prostate cancer. To answer this question, men who have chosen prostatectomy will be randomly assigned to preoperative treatment with celecoxib or placebo for four weeks. Carefully collected tumor, premalignant, and benign prostate tissue will then be examined for apoptosis, androgen receptor and prostaglandin E2 levels. Tumor COX-2 expression will be correlated with observed treatment effects. The data generated by this study will serve as a foundation for the development of COX-2 targeted therapies for prostate cancer, will provide preliminary evidence for larger scale clinical trials aimed at treatment and prevention of prostate cancer, and will validate current preclinical models used to study COX-2 in prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

I. To determine if COX-2 inhibition with celecoxib significantly increases apoptosis in human adenocarcinoma of the prostate.

SECONDARY OBJECTIVES

I. To determine if COX-2 inhibition with celecoxib reduces levels of Prostaglandin E2 and androgen receptor in fresh tumor tissue collected at prostatectomy

II. To collect pre- and postoperative serum Prostate Specific Antigen (PSA) for exploratory analyses

III. To determine the effect of celecoxib on adverse effects, perioperative surgical complications and post surgery analgesic use

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically proven adenocarcinoma of the prostate and planned prostatectomy
* Age >= 18
* Performance status (ECOG <= 2)
* Hemoglobin > 10 g/dL (within 4 weeks)
* Creatinine <= 1.5 mg/dL
* Signed informed patient consent

Exclusion Criteria:

* Other preoperative or prior treatment directed at prostate cancer
* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* Use of non-steroidal anti-inflammatory agents within seven days of celecoxib treatment
* Hypersensitivity to celecoxib
* A history of asthma, urticaria, or anaphylaxis precipitated by an NSAID
* History of significant upper gastrointestinal bleeding or active peptic ulcer disease
* Current treatment with anticoagulants
* Allergy to sulfonamide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Apoptosis Index, defined as the percent positive staining cells | approximately 4 weeks of treatment
  Percent positively staining cells with a minimum of 1000 total cells counted. Descriptive statistics will be conducted. The apoptotic index will be reported with 95% confidence intervals.

SECONDARY OUTCOMES:
Prostaglandin and Androgen Receptor Levels | approximately 4 weeks of treatment
  Descriptive statistical analysis will be conducted. The estimates will be reported with 95% confidence intervals.
Percent Change in Median PSA Values, pre- and postoperatively | approximately 4 weeks of treatment
  Pre- and postoperative PSA will be collected. Descriptive statistics will be conducted, comparing preoperative PSA level to postoperative level.
Perioperative Analgesic Use, using morphine equivalents | Prostatectomy to discharge from hospital, no more than 30 days post prostatectomy
  Descriptive statistical analysis will be conducted. The estimate will be calculated using morphine equivalents dividend by length of hospital stay and reported with 95% confidence intervals.
Surgical Complications, defined as incidence of adverse events determined to be related to surgery graded by NCI CTCAE version 2.0 | Intraoperatively to 30 days postoperatively
  Intraoperative and post surgical complications will be collected and reported.
Incidence of Adverse Events, graded by NCI CTCAE version 2.0 | From start of treatment to 30 days post prostatectomy
  Descriptive statistical analysis will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M Beer, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon